CLINICAL TRIAL: NCT07307170
Title: The Analgesic Efficacy and Safety of Oral Medications (Mirogabalin) in Patients With Herpes Zoster
Brief Title: The Analgesic Efficacy and Safety of Mirogabalin in Patients With Herpes Zoster
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Fang Luo, Director, Department of Pain Management, Principal Investigator, Clinical Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-369-02-1
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Herpes Zoster; Mirogabalin; Pain
MeSH Terms: conditions — Herpes Zoster; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirogabalin group (Experimental)
  Interventions: Drug: Mirogabalin combined conventional therapy
- Control group (Active Comparator)
  Interventions: Drug: Conventional therapy

INTERVENTIONS:
Drug: Mirogabalin combined conventional therapy — In the mirogabalin combined conventional therapy group, mirogabalin will be initiated at 5 mg twice daily. After at least one week, the dose will be increased by 5 mg each time based on individual patient response and tolerability, until a dose of 15 mg twice daily reached, with a maximum dose of 15 mg twice daily. In addition, the group will contain conventional treatment for HZ, except mirogabalin, including NSAIDs, opioids, antiviral drugs and so on.
  Arms: Mirogabalin group
Drug: Conventional therapy — In the conventional therapy group, treatments will include NSAIDs, opioids, antiviral drugs and so on.
  Arms: Control group

SUMMARY:
Herpes zoster (HZ) is characterized by a painful dermatomal rash and significantly affects quality of life, with acute pain increasing the risk of postherpetic neuralgia. Although early antiviral therapy limits viral replication, its analgesic effect is insufficient, and many patients experience inadequate relief despite stepwise use of non-opioids and opioids. Gabapentinoids such as gabapentin and pregabalin are recommended adjuncts, but their efficacy in acute HZ is inconsistent and often accompanied by adverse effects that limit tolerability. Mirogabalin, a newer gabapentinoid approved for peripheral neuropathic pain, has higher affinity and slower dissociation from the α2δ-1 subunit, suggesting stronger analgesia with fewer central side effects. However, its role in managing acute HZ pain remains unknown. We therefore hypothesize that adding mirogabalin to conventional therapy will provide superior pain relief compared with standard treatment alone, and propose a prospective, randomized, controlled, open-label, blinded-endpoint trial to evaluate this.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ages more than 18 years;
* 2. Patients with onset of HZ rash less than 90 days;
* 3. Experiencing moderate to severe HZ pain with an average pain score of at least 4 on a Numeric Rating Scale (NRS, 0 = no pain, 10 = worst possible pain);
* 4. Aspartate aminotransferase and alanine aminotransferase levels less than twice the upper limit of normal;
* 5. Estimated glomerular filtration rate of 30 mL/min per 1.73 m2 or higher;
* 6. Willing to sign the informed consent form and possessing sufficient cognitive and language abilities to comply with all the study requirements.

Exclusion Criteria:

* 1. History of taking gabapentin or pregabalin;
* 2. Patients with evidence of cutaneous or visceral dissemination of HZ infection (cutaneous dissemination is defined as more than 20 discrete lesions outside adjacent dermatomes) or ocular involvement of HZ;
* 3. History of intolerance or hypersensitivity to any active components or excipient of the mirogabalin;
* 4. History of systemic immune diseases, organ transplantation, or cancers;
* 5. Pregnancy or breastfeeding;
* 6. Suffering from acute or chronic pain disorders other than HZ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
the average numeric rating scale score over the past 24 hours, rated each morning upon awakening and average over 7 days at week 4 | At week 4 after experimental drug medication
  The numeric rating scale (NRS) score is a way to quantify the degree of subjective feelings such as pain using numbers. Generally, 0 represents no pain, and 10 represents the most severe pain. A higher score indicates more severe pain.

SECONDARY OUTCOMES:
The worst numeric rating scale score | at weeks 1, 2, 4, 8, and 12 after experimental drug medication
  The numeric rating scale (NRS) score is a way to quantify the degree of subjective feelings such as pain using numbers. Generally, 0 represents no pain, and 10 represents the most severe pain. A higher score indicates more severe pain.
Proportion of Patients Achieving Pain Reduction | at weeks 1, 2, 4, 8, and 12 after experimental drug medication
  The proportion of patients achieving a ≥ 50% and ≥ 30% reduction in mean baseline pain intensity
Proportion of patients developing postherpetic neuralgia | at week 12 after experimental drug medication
The type of analgesics and average weekly consumption per analgesics | at weeks 4, 8, and 12 after experimental drug medication
The 12-item Short-Form Health Survey (SF-12) score | at weeks 4, 8, and 12 after experimental drug medication
  The SF-12 score assesses the health-related quality of life, capturing preferences across various health states. It assesses 8 dimensions: physical functioning, physical role limitations due to physical health, bodily pain, general health, vitality, social functioning, emotional role limitations due to emotional problems, and mental health. Scores range from 0 to 100 for each dimension, with higher scores indicating better health status.
The Medical Outcomes Study Sleep Scale (MOS) | at weeks 4, 8, and 12 after experimental drug medication
  The MOS is a questionnaire comprising 12 items that assess various aspects of sleep using a 6-point ordinal scale (1 indicating permanence and 6 indicating absence).
Adverse events | Through study completion, an average of 12 weeks
  The incidence and proportion of AEs will be recorded and categorized as mild, moderate, severe, or life-threatening. AEs are defined as events that arise during treatment, were absent before treatment, or worsen relative to the pretreatment state.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing 100070, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures and appendices) are available. Derived data supporting the findings of this study are available from the corresponding author Fang Luo on request.

REFERENCES:
- See also: Rosamilia LL. Herpes Zoster Presentation, Management, and Prevention: A Modern Case-Based Review. Am J Clin Dermatol. 2020;21(1):97-107. — https://pubmed.ncbi.nlm.nih.gov/31741185/
- See also: Liu Y, Xiao S, Li J, Long X, Zhang Y, Li X. A Network Meta-Analysis of Randomized Clinical Trials to Assess the Efficacy and Safety of Antiviral Agents for Immunocompetent Patients with Herpes Zoster-Associated Pain. Pain Physician. 2023;26(4):337-46. — https://pubmed.ncbi.nlm.nih.gov/37535772/
- See also: Domon Y, Arakawa N, Inoue T, Matsuda F, Takahashi M, Yamamura N, et al. Binding Characteristics and Analgesic Effects of Mirogabalin, a Novel Ligand for the α2δ Subunit of Voltage-Gated Calcium Channels. J Pharmacol Exp Ther. 2018;365(3):573-82. — https://pubmed.ncbi.nlm.nih.gov/29563324/